CLINICAL TRIAL: NCT01114932
Title: The Optimum Time for Preoxygenation Based on Body Mass Index
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Residency program director, Department of anesthesiology, Cedars-Sinai Medical Center
Other Study IDs: Pro00011544
Record Dates: First submitted 2010-04-23; First posted 2010-05-03 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Body Weight; Obesity
Keywords: pre-oxygenation; body mass index; end-tidal O2; anesthesia induction
MeSH Terms: conditions — Body Weight; Obesity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- BMI-I: Patients with BMI values between 18.5-24.9
- BMI-II: Patients with BMI values between 25-29.9
- BMI-III: Patients with BMI values between 30-49.9

SUMMARY:
The purpose of this study is to evaluate the relationship between the time needed to raise the oxygen concentration in patient's blood to 90% and his/or her body mass index. The prevalence of obesity in our society continues to rise. No studies have shown the time required for preoxygenation (oxygen given) in relation to body mass index (body weight in kg/height in meter2).

DETAILED DESCRIPTION:
100% oxygen given to patient before induction of anesthesia (asleep) is the standard clinical care. However, studies using various methods have shown differences in terms of the optimal time, technique and number of breaths needed for efficient oxygenation. The only difference to the standard pre-anesthesia care is that we will record the time to raise patient oxygen to 90%. Age is recorded to ensure that the subjects fall within our inclusion criteria. The weight (W) in kilograms and height (H) in meters will be used to calculate the body mass index (BMI): BMI = W/H2. Alveolar oxygen uptake is dependent on respiratory rate, heart rate, blood pressure, temperature and hemoglobin level. These parameters are measured in order to identify factors that may affect the accuracy of the study. We will record the pulse oximetry value to note the initial oxygen saturation on room air and after the oxygenation.

Facial hair and mask fit are recorded to assess possible failure of an optimal facemask seal. End-tidal carbon dioxide (FE'CO2) is also measured to ensure an adequate facemask seal. Anxiety can increase the respiratory rate, heart rate and affect patient compliance with a fitted facemask. All of the aforementioned values are recorded to assess reasons for possible failure of the preoxygenation technique and inaccurate results.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 18-50 years with no limitations as to gender or race
* Participants classified as ASA 1 or 2
* Participants capable of understanding and signing an informed consent

Exclusion Criteria:

* Conditions which would affect their oxygenation such as heart disease, lung disease, anemia (Hemoglobin less than 12 g/dL)
* History of smoking (smoking can affect pulmonary function and oxygen carrying capacity)
* Acute substance abuse (substance abuse can affect respiratory function).
* Maxillofacial abnormalities which would interfere with proper face mask seal.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of 100 subjects between the ages of 18-50 classified as ASA 1 or 2 with no limitations as to gender or race that are scheduled for elective surgery at Cedars-Sinai Medical Center. There are changes to lung functioning as functional residual capacity (FRC), closing capacity, and lung volume after age 50; therefore, the age limitation is set to age 50. Changes in lung and chest wall compliance necessitate the exclusion of anyone over the age of 50. Minors are also excluded as there is difficulty fitting the face mask due to a smaller physiology.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2007-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Time to reach 90% end tidal oxygen saturation using monitor and stop watch | 1 to 10 minutes
  Using monitors on the anesthesia machine, we recorded the end tidal oxygen saturation value and also recorded the time at which the end tidal oxygen was recorded. From the information collected the relationship between BMI and gender with the time to 90% end tidal oxygen saturation will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States